CLINICAL TRIAL: NCT04313088
Title: Double Blind, Placebo Controlled, Cross Over Study to Investigate the Effectiveness and Safety of Eluxadoline in the Treatment of Diabetic Diarrhea
Brief Title: Investigation of Eluxadoline for Diabetic Diarrhea
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: This study did not enroll any subjects
Sponsor: Temple University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 26347
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Diabetic Diarrhea; Diabetes; Diarrhea
Keywords: eluxadoline; Viberzi
MeSH Terms: conditions — Diabetes Mellitus; Diarrhea | interventions — eluxadoline

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized 1:1 via random number generator to either receive eluxadoline 100mg twice daily (BID) or matching placebo. Participants will take assigned medication or placebo as prescribed for 42 days. A washout phase will take place on days 43-70. On days 71-112, participants will crossover and take either eluxadoline 100mg BID or matching placebo based on their previously assigned group. Throughout the study, weekly phone calls with a study coordinator will take place and participants will keep a daily stool diary. Office visits with a physician will take place at the beginning of the pre-randomization phase and at Day 0, 42, 70 and 112 of the study phase. Participants will refrain from use of all additional anti-diarrheal medication during the entirety of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization assignments will be handled by the statistician by means of a random number generator and assignments will be kept in opaque envelopes. The randomization scheme will be passed to the Temple Pharmacist. Based on the number, the Temple Pharmacist will dispense directly to the patient either drug or placebo in a labeled, child proof, pill bottle in a manner that does not disclose which group the patient is assigned. The Temple Pharmacist that is not a participant in the study will be responsible for dispensing study medication and will keep a secured log with the identity of that which is dispensed in case un-blinding becomes necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group A (Other): All eligible patients will receive both eluxadoline and placebo, however each patient will be randomized to the order in which this happens. Eligible patients will be randomized 1:1 via random number generator to either receive eluxadoline 100mg twice daily then matching placebo or placebo then eluxadoline 100mg twice daily. Participants in Group A will take eluxadoline 100mg by mouth twice for 42 days. A washout phase will take place on days 43-70 where no study drug or placebo will be administered. On days 71-112, participants will crossover and take matching placebo by mouth twice daily. Each participant in Group A will take 42 days of eluxadoline 100mg twice daily followed by 42 days of placebo over the course the study.
  Interventions: Drug: Eluxadoline 100 mg
- Experimental Group B (Other): All eligible patients will receive both eluxadoline and placebo, however each patient will be randomized to the order in which this happens. Eligible patients will be randomized 1:1 via random number generator to either receive eluxadoline 100mg twice daily then matching placebo or placebo then eluxadoline 100mg twice daily. Participants in Group B will take placebo by mouth twice daily for 42 days. A washout phase will take place on days 43-70 where no study drug or placebo will be administered. On days 71-112, participants will crossover and take eluxadoline 100mg by mouth twice daily. Each participant in Group B will take 42 days of placebo followed by 42 days of eluxadoline 100mg twice daily over the course the study.
  Interventions: Drug: Eluxadoline 100 mg

INTERVENTIONS:
Drug: Eluxadoline 100 mg — Eluxadoline 100mg by mouth twice daily with food
  Other Names: Viberzi

SUMMARY:
Diabetes is a chronic disease that affects a large part of the United States population. The majority of patients with diabetes will experience gastrointestinal symptoms. One of the most troublesome gastrointestinal symptoms that diabetes can cause is diarrhea, otherwise known as "Diabetic Diarrhea." This occurs because diabetes does damage to nerves that control the gut and prevent it from functioning normally. Currently, there are only several medications used to treat the symptoms of Diabetic Diarrhea, but many of these medications have serious side effects or do not work well.

We are investigating the drug eluxadoline for the treatment of Diabetic Diarrhea. Eluxadoline is a gut-specific medication that is FDA approved to treat diarrhea related to irritable bowel syndrome (IBS-D). Our hypothesis is eluxadoline will safely and successfully reduce diarrhea symptoms (number of stools and less liquid stools) and improve the quality of life in patients with Diabetic Diarrhea when compared with placebo. Each patient with Diabetic Diarrhea who participates will take both eluxadoline and a placebo drug at separate times over a period of several months as part of a crossover study design. While on each medication, eluxadoline or placebo, the participants will keep a diary of symptoms and will be followed by the medical team through a combination of office visits and questionnaires. There will be five planned office visits and intermittent phone calls (questionnaires, surveys) over the 140-day study period. Participants will not be permitted to use any other anti-diarrhea medication during the study period and will continue on medication for management of their diabetes.

DETAILED DESCRIPTION:
Over 30 million Americans have been diagnosed with diabetes and the related complications account for the 7th most common cause of death in the United States. Within the gastrointestinal system, diabetic enteropathy can manifest in a variety of ways of which diarrhea (DD) may be amongst the most debilitating. The prevalence of DD has been estimated to approach 20%. Autonomic neuropathy, loss of nitrergic neurons and loss of stimulation of alpha adrenergic neurons have all been postulated to have an effect on gut motility and water reabsorption. New research may indicate that chronic hyperglycemia damages Interstitial Cells of Cajal and other enteric nerves through oxidative stress to cause symptoms. Other areas of emerging research have explored the role of enteric hormones, smooth muscle cell abnormalities, inflammatory mediators, enteric glial cells, and the patients' microbiome as factors in the pathogenesis of DD Globally, symptoms of DD are inversely correlated with glycemic control. DD is a diagnosis of exclusion and its associated voluminous, watery stools are often unresponsive to conventional therapy.

Eluxadoline has emerged as an FDA approved drug for the treatment of IBS-D. It is an agonist of mu and kappa opioid receptors while also an antagonist at delta receptors in the gut. Through these mechanisms, eluxadoline acts to slow peristalsis while at the same time prevents constipation and provides pain relief to patients with IBS-D. Given its success in the treatment of IBS-D, we hypothesize that eluxadoline will safely bring significant symptom relief and improve quality of life for patients with DD.

Our study is a double blind, placebo controlled cross over design to investigate the safety and effectiveness of eluxadoline in relieving the symptoms of DD. Diabetic patients over the age of 18 with diarrhea for which an alternative underlying etiology has not been identified will be eligible to participate in a pre-randomization phase lasting four weeks to document baseline symptoms. At the conclusion of the pre-randomization period, patients will be randomized to either Experimental Group A or Experimental Group B. Randomization will be performed by a statistician and only the Temple Pharmacist will be aware of the group assignment to distribute study drug or placebo. Participants will receive either eluxadoline 100mg by mouth twice daily or matching placebo for 42 days, complete a washout period of 28 days when neither placebo or eluxadoline will be given, and then continue on by taking either eluxadoline or placebo for an additional 42 days based on which experimental group they have been assigned. Throughout the study period, patients will keep a daily stool diary, participate in questionnaires administered by a study coordinator and have pre-determined follow up office visits with study physicians.

The primary endpoint compared between eluxadoline and placebo will be proportion of days in which all bowel movements for that day have a consistency on the Bristol Stool Scale <5. Secondary endpoints will be improvement on the subject's Likert scores for global satisfaction, score on the Diabetes-39 and Facit-D questionnaires as well as proportion of days with fecal incontinence and nights with nocturnal diarrhea. We hypothesize that compared to placebo, eluxadoline will significantly improve the primary and secondary endpoints described above.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Documented diabetes mellitus (DM) Type I or DM Type II - must be on medical therapy
* ≥ 3 bowel movements per day with Bristol type 6 or 7 stools at least 4 days per week for > 6 months. They must continue to meet these criteria during the 4 week pre-randomization phase.
* Normal sigmoidoscopy or colonoscopy with biopsies negative for microscopic colitis
* Negative work up for Clostridium difficile
* Negative work up for Celiac Disease either by assessment of serum tissue transglutaminase Immunoglobulin A (IgA) or by small bowel biopsy
* Normal fecal elastase and fecal calprotectin levels
* Normal thryoid stimulating hormone (TSH) level

Exclusion Criteria:

* Subjects who, in the estimation of the investigator, have drug-induced diarrhea
* Subjects unwilling to stop anti-diarrheal medications during the study
* Pregnancy or nursing mothers
* History of Cholecystectomy or Sphincter of Oddi Dysfunction
* Patients unable to undergo sigmoidoscopy or colonoscopy
* Patients with a history of inflammatory bowel disease (IBD)
* Prior history of pancreatitis
* Patients with hepatic impairment
* Patients who consume ≥ 3 alcoholic beverages per day
* Patients on oral opioids, who abuse illicit opioids, or have had a history of opioid abuse
* Patients on OATP1B1 Inhibitors (Rifampicin, Clarithromycin, Erythromycin, Cyclosporine, Gemfibrozil)
* Patients for whom inclusion in the study would be dangerous
* Subjects unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of days with improved bowel movements | 140 days
  Proportion of days in which all recorded bowel movements for that day have a consistency on the Bristol Stool Scale of < 5.
  Scale:
  Type 1: Separate hard lumps, like nuts (hard to pass) Type 2: Sausage-shaped, but lumpy Type 3: Like a sausage but with cracks on its surface Type 4: Like a sausage or snake, smooth and soft Type 5: Soft blobs with clear cut edges (easy to pass) Type 6: Fluffy pieces with ragged edges, a mushy stool Type 7: Watery, no solid pieces, entirely liquid

SECONDARY OUTCOMES:
Likert score for global satisfaction | 140 days
  > 1 point improvement in the subject's Likert scores for global satisfaction with treatment
  Scale:
  High score means higher satisfaction
  1. - Strongly disagree
  2. - Disagree
  3. - Somewhat disagree
  4. - Neither agree nor disagree
  5. - Somewhat agree
  6. - Agree
  7. - Strongly agree
Diabetes quality of life | 140 days
  Score on the Diabetes-39 (DM QoL questionnaire)
  Scale:
  1 - 7, with 1 being "not affected at all" and 7 being "extremely affected"
Diarrhea quality of life | 140 days
  Score on the Facit-D (v. 4.0) - QoL questionnaire specific for diarrhea
  Scale:
  0 - Not at all
  1. - A little bit
  2. - Somewhat
  3. - Quite a bit
  4. - Very much
Fecal incontinence | 140 days
  Proportion of days with fecal incontinence
Nocturnal diarrhea | 140 days
  Proportion of days with nocturnal diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Reichenbach, MD,PhD, Principal Investigator — Lewis Katz School of Medicine at Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gotfried J, Priest S, Schey R. Diabetes and the Small Intestine. Curr Treat Options Gastroenterol. 2017 Dec;15(4):490-507. doi: 10.1007/s11938-017-0155-x. PMID 28913777
- [Background] Mourad FH, Gorard D, Thillainayagam AV, Colin-Jones D, Farthing MJ. Effective treatment of diabetic diarrhoea with somatostatin analogue, octreotide. Gut. 1992 Nov;33(11):1578-80. doi: 10.1136/gut.33.11.1578. PMID 1452087
- [Background] Bytzer P, Talley NJ, Leemon M, Young LJ, Jones MP, Horowitz M. Prevalence of gastrointestinal symptoms associated with diabetes mellitus: a population-based survey of 15,000 adults. Arch Intern Med. 2001 Sep 10;161(16):1989-96. doi: 10.1001/archinte.161.16.1989. PMID 11525701
- [Background] Camilleri M, Malagelada JR. Abnormal intestinal motility in diabetics with the gastroparesis syndrome. Eur J Clin Invest. 1984 Dec;14(6):420-7. doi: 10.1111/j.1365-2362.1984.tb01206.x. PMID 6441717
- [Background] Yoneda S, Kadowaki M, Kuramoto H, Fukui H, Takaki M. Enhanced colonic peristalsis by impairment of nitrergic enteric neurons in spontaneously diabetic rats. Auton Neurosci. 2001 Sep 17;92(1-2):65-71. doi: 10.1016/S1566-0702(01)00317-4. PMID 11570705
- [Background] Yagihashi S, Sima AA. Diabetic autonomic neuropathy in BB rat. Ultrastructural and morphometric changes in parasympathetic nerves. Diabetes. 1986 Jul;35(7):733-43. doi: 10.2337/diab.35.7.733. PMID 3721060
- [Background] Yagihashi S, Sima AA. Neuroaxonal and dendritic dystrophy in diabetic autonomic neuropathy. Classification and topographic distribution in the BB-rat. J Neuropathol Exp Neurol. 1986 Sep;45(5):545-65. doi: 10.1097/00005072-198609000-00005. PMID 3746344
- [Background] Chandrasekharan B, Anitha M, Blatt R, Shahnavaz N, Kooby D, Staley C, Mwangi S, Jones DP, Sitaraman SV, Srinivasan S. Colonic motor dysfunction in human diabetes is associated with enteric neuronal loss and increased oxidative stress. Neurogastroenterol Motil. 2011 Feb;23(2):131-8, e26. doi: 10.1111/j.1365-2982.2010.01611.x. Epub 2010 Oct 12. PMID 20939847
- [Background] Yarandi SS, Srinivasan S. Diabetic gastrointestinal motility disorders and the role of enteric nervous system: current status and future directions. Neurogastroenterol Motil. 2014 May;26(5):611-24. doi: 10.1111/nmo.12330. Epub 2014 Mar 24. PMID 24661628
- [Background] D'Addio F, Fiorina P. Type 1 Diabetes and Dysfunctional Intestinal Homeostasis. Trends Endocrinol Metab. 2016 Jul;27(7):493-503. doi: 10.1016/j.tem.2016.04.005. Epub 2016 May 13. PMID 27185326
- [Background] Zanoni JN, Buttow NC, Bazotte RB, Miranda Neto MH. Evaluation of the population of NADPH-diaphorase-stained and myosin-V myenteric neurons in the ileum of chronically streptozotocin-diabetic rats treated with ascorbic acid. Auton Neurosci. 2003 Feb 28;104(1):32-8. doi: 10.1016/S1566-0702(02)00266-7. PMID 12559201
- [Background] Izbeki F, Wittman T, Rosztoczy A, Linke N, Bodi N, Fekete E, Bagyanszki M. Immediate insulin treatment prevents gut motility alterations and loss of nitrergic neurons in the ileum and colon of rats with streptozotocin-induced diabetes. Diabetes Res Clin Pract. 2008 May;80(2):192-8. doi: 10.1016/j.diabres.2007.12.013. Epub 2008 Feb 1. PMID 18242757
- [Background] Chang EB, Bergenstal RM, Field M. Diarrhea in streptozocin-treated rats. Loss of adrenergic regulation of intestinal fluid and electrolyte transport. J Clin Invest. 1985 May;75(5):1666-70. doi: 10.1172/JCI111874. PMID 2987308
- [Background] He CL, Soffer EE, Ferris CD, Walsh RM, Szurszewski JH, Farrugia G. Loss of interstitial cells of cajal and inhibitory innervation in insulin-dependent diabetes. Gastroenterology. 2001 Aug;121(2):427-34. doi: 10.1053/gast.2001.26264. PMID 11487552
- [Background] Luo P, Liu D, Li C, He WX, Zhang CL, Chang MJ. Enteric glial cell activation protects enteric neurons from damage due to diabetes in part via the promotion of neurotrophic factor release. Neurogastroenterol Motil. 2018 Oct;30(10):e13368. doi: 10.1111/nmo.13368. Epub 2018 May 8. PMID 29740907
- [Background] Fant RV, Henningfield JE, Cash BD, Dove LS, Covington PS. Eluxadoline Demonstrates a Lack of Abuse Potential in Phase 2 and 3 Studies of Patients With Irritable Bowel Syndrome With Diarrhea. Clin Gastroenterol Hepatol. 2017 Jul;15(7):1021-1029.e6. doi: 10.1016/j.cgh.2017.01.026. Epub 2017 Feb 3. PMID 28167156
- [Background] Munjal A, Dedania B, Cash B. Update on Pharmacotherapy for Irritable Bowel Syndrome. Curr Gastroenterol Rep. 2019 Apr 25;21(6):25. doi: 10.1007/s11894-019-0692-7. PMID 31025114
- [Background] Chen Y, Liu G, He F, Zhang L, Yang K, Yu H, Zhou J, Gan H. MicroRNA 375 modulates hyperglycemia-induced enteric glial cell apoptosis and Diabetes-induced gastrointestinal dysfunction by targeting Pdk1 and repressing PI3K/Akt pathway. Sci Rep. 2018 Aug 23;8(1):12681. doi: 10.1038/s41598-018-30714-0. PMID 30140011
- [Background] Bodi N, Szalai Z, Bagyanszki M. Nitrergic Enteric Neurons in Health and Disease-Focus on Animal Models. Int J Mol Sci. 2019 Apr 24;20(8):2003. doi: 10.3390/ijms20082003. PMID 31022832
- [Background] Selby A, Reichenbach ZW, Piech G, Friedenberg FK. Pathophysiology, Differential Diagnosis, and Treatment of Diabetic Diarrhea. Dig Dis Sci. 2019 Dec;64(12):3385-3393. doi: 10.1007/s10620-019-05846-6. No abstract available. PMID 31541370